CLINICAL TRIAL: NCT06907927
Title: Using Artificial Intelligence to Improve Radiologists' Performance in Radiology Report Writing: a Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-0033
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Behavioral: Control group
- Experimental group (Experimental)
  Interventions: Behavioral: Experimental group

INTERVENTIONS:
Behavioral: Control group — the radiologists enrolled in the study will be randomly divided into two groups: the experimental group used AI(Artificial Intelligence) software to assist in the submission of radiology reports and the control group did not use any AI software to submit their reports
  Arms: Control group
Behavioral: Experimental group — the radiologists enrolled in the study will be randomly divided into two groups: the experimental group used AI(Artificial Intelligence) software to assist in the submission of radiology reports and the control group did not use any AI software to submit their reports
  Arms: Experimental group

SUMMARY:
This is a randomised controlled trial to assess whether artificial intelligence software can improve radiologists' performance in radiology report writing and improve the quality of radiology reports.

ELIGIBILITY:
Inclusion Criteria:

1. Radiologists who submit reports;
2. Clinical experience of less than 10 years and more than six months;
3. An average of more than 10 radiology reports are submitted per day;
4. Participants provided signed informed consent.

Exclusion criteria：

1. Radiologists who review reports;
2. Clinical experience of less than 6 months or more than 10 years;
3. An average of less than 10 radiology reports are submitted per day.）

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Error rates in radiology reports | 1 month
  Statistical analysis of errors in radiology reports submitted by study and control group physicians

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China